CLINICAL TRIAL: NCT06686030
Title: An Exploratory, Multi-cohort Phase II Study of Combination Therapy of AK112 With Chemotherapy and/or Olaparib in Platinum-sensitive Ovarian Cancer
Brief Title: Combination Therapy of AK112 With Chemotherapy and/or Olaparib in Platinum-sensitive Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK112-211
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Platinum-sensitive Ovarian Cancer
Keywords: platinum-sensitive ovarian cancer; PD-1; VEGF; antibody; AK112
MeSH Terms: interventions — Drug Therapy; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1-10 (BRCAm) (Experimental): AK112(10mg/kg)+chemo for 4-6 cycles, AK112 (10mg/kg)+Olaparib maintenance
  Interventions: Drug: AK112 low dose; Drug: Chemotherapy; Drug: Olaparib
- Cohort 1-10B (non-BRCAm) (Experimental): AK112(10mg/kg)+chemo for 4-6cycles, AK112(10mg/kg) maintenance
  Interventions: Drug: AK112 low dose; Drug: Chemotherapy
- Cohort 1-20A (BRCAm) (Experimental): AK112(20mg/kg)+chemo for 4-6cycles, AK112(20mg/kg)+Olaparib maintenance
  Interventions: Drug: Chemotherapy; Drug: Olaparib; Drug: AK112 high dose
- Cohort 1-20B (non-BRCAm) (Experimental): AK112(20mg/kg)+chemo for 4-6cycles, AK112(20mg/kg) maintenance
  Interventions: Drug: Chemotherapy; Drug: AK112 high dose
- Cohort 2 (Prior ≥2L) (Experimental): AK112(20mg/kg)+Olaparib
  Interventions: Drug: Olaparib; Drug: AK112 high dose

INTERVENTIONS:
Drug: AK112 low dose — 10mg/kg, Q3W, ivgtt
  Other Names: Ivonescimab
  Arms: Cohort 1-10 (BRCAm); Cohort 1-10B (non-BRCAm)
Drug: Chemotherapy — ivgtt
  Arms: Cohort 1-10 (BRCAm); Cohort 1-10B (non-BRCAm); Cohort 1-20A (BRCAm); Cohort 1-20B (non-BRCAm)
Drug: Olaparib — bid, oral
  Arms: Cohort 1-10 (BRCAm); Cohort 1-20A (BRCAm); Cohort 2 (Prior ≥2L)
Drug: AK112 high dose — 20mg/kg, Q3W, ivgtt
  Arms: Cohort 1-20A (BRCAm); Cohort 1-20B (non-BRCAm); Cohort 2 (Prior ≥2L)

SUMMARY:
An Exploratory, Multi-cohort Phase II Study of combination therapy of AK112 with chemotherapy and/or olaparib in platinum-sensitive ovarian cancer(PSOC)

DETAILED DESCRIPTION:
This is a Phase 2, open label, multicohort, multicenter study designed to evaluate the efficacy and safety of combination of AK112 with chemotherapy and/or olaparib in platinum-sensitive ovarian cancer. AK112 is a bispecific monoclonal antibody targeting VEGF and PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. Signs the written informed consent form.
2. Female participants who are at least 18 years of age on the day of signing informed consent with.
3. ECOG of 0 or 1.
4. Life expectancy ≥3 months.
5. Histologically documented epithelial and non-mucinous PSOC. PSOC was defined as radiographic progression greater than 6 months from last dose of platinum-based chemotherapy.

   Note:
   1. If breast cancer susceptibility gene (BRCA) positive participants must have received prior treatment with a poly adenosine phosphate-ribose polymerase inhibitor (PARPi).
   2. Ovarian cancer includes ovarian cancer, fallopian tube cancer and primary peritoneal cancer in this study, unless otherwise specified.
6. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team.
7. Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue.
8. Has adequate organ function.
9. All subjects of reproductive potential must agree to use an effective method of contraception, during and for 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Other pathological types such as mucinous cancer, sex cord stromal cell tumor, etc.
2. Presence of central nervous system (CNS) metastases or carcinomatous meningitis.
3. Subjects with uncontrollable pleural, pericardial, or peritoneal effusion requiring repeated drainage.
4. Subjects with other active malignancies within 3 years prior to randomization.
5. Received systemic anti-tumor therapy within 2 weeks prior to randomization.
6. Any prior treatments targeting the mechanism of tumor immunity.
7. Major surgical , open biopsy or significant trauma within 4 weeks prior to randomization; or elective major surgical treatment required during the study.
8. Active or potentially recurrent autoimmune disease.
9. Subjects who require systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to randomization.
10. Receiving live vaccines within 4 weeks prior to randomization.
11. Known primary or secondary immunodeficiencies, including testing positive for human immunodeficiency virus (HIV) antibodies.
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Known history of interstitial lung disease or non-infectious pneumonitis.
14. Serious infections requiring hospitalization.
15. Presence of active infection requiring systemic therapy.
16. Subjects with active hepatitis B and active viral hepatitis C.
17. Active or documented inflammatory bowel diseases, active diverticulitis.
18. Subjects with clinically significant cardio-cerebrovascular disease.
19. Unresolved toxicities from prior anticancer therapy.
20. History of severe hypersensitivity reactions to other mAbs.
21. Pregnant or lactating women.
22. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug.
23. Exclusion Criteria for combination therapy-Related: For cohort 1: Known contraindications or allergy to paclitaxel or carboplatin. For Cohorts 1-10A, Cohort 1-20A, and Cohort 2: Known contraindications or allergy to Olaparib.
24. Exclusion Criteria for AK112-Related: Known contraindications or allergy to any component of VEGF mABs or any medical conditions that affect the safety of AK112.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by investigator per RECIST v1.1 | up to 2 years
  PFS is defined as the time from the date of first dosing till the first documented disease progression Per RECIST v1.1 assessed by the investigator or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by investigator | Up to 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Disease control rate(DCR)assessed by investigator per RECIST v1.1 | Up to 2 years
  Proportion of subjects who have received response(ie complete response or partial response) or stable disease relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Duration of Response (DOR) assessed by investigator per RECIST v1.1 | Up to 2 years
  DOR means time measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Time to Response (TTR) assessed by investigator per RECIST v1.1 | Up to 2 years
  TTR refers to Time to Response.
Overall Survival(OS) | Up to 2 years
  OS is defined as the time from randomization or first dosing to death due to any cause.
Number of participants with adverse event (AE) | Up to 2 years
  The number of participants experiencing an AE and the severity of AEs will be assessed. AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science And Technology, Wuhan, China